CLINICAL TRIAL: NCT04363749
Title: Do Respiratory Control Center Anomalies Explain the Lack of Respiratory Sensations Perceptions Observed in Patients Affected by COVID-19 ?
Brief Title: COVID-19 Infection: Exploration of Respiratory Control Center Abnormalities
Acronym: CRC-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP200476
Record Dates: First submitted 2020-04-20; First posted 2020-04-27 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Neurological Complication
Keywords: SARS-CoV-2; COVID-19; dyspnea; hypoxic stimulus
MeSH Terms: conditions — COVID-19; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15 COVID positive patients (Experimental): dyspnea rating to various dyspneic stimulus
  Interventions: Other: hypoxia : 14.3 and 12.7% FIO2, hypercapnia 7% CO2, inspiratory mechanical constraint
- 15 healthy controls (Active Comparator): dyspnea rating to various dyspneic stimulus
  Interventions: Other: hypoxia : 14.3 and 12.7% FIO2, hypercapnia 7% CO2, inspiratory mechanical constraint

INTERVENTIONS:
Other: hypoxia : 14.3 and 12.7% FIO2, hypercapnia 7% CO2, inspiratory mechanical constraint — the fraction of inspired oxygen is reduced from ~21% (room air) to 14.3 and 12.7% allowing the SpO2 to decrease to ~75%, rebreathing test allowing the PCO2 to rise to 65 mmHg, inspiratory mechanical constraint with 50 to 75% of maximum inspiratory pressure

SUMMARY:
The purpose of the present study is to determine whether there is a decrease in the emotional response to experimental induction of dyspnea by hypoxic stimulation in subjects with a "neurological" form of COVID-19, compared to healthy controls.

DETAILED DESCRIPTION:
SARS CoV-2 infection causes lung damage that can be severe enough to require artificial ventilation. Clinicians taking care of these patients are surprised by the scant respiratory sensations and emotional responses described by patients. This attenuation of respiratory interoception deprives clinicians of the usual warning signs during respiratory decompensation of dyspnea and its aggravation. It may be the result of central nerve damage. This hypothesis is bolstered by the observation that within the multiple clinical forms of COVID-19 infection there are some "neurological" forms (headache, anosmia, agueusia, dizziness, without respiratory signs and with little or no fever), that are most likely the consequence of olfactory penetration of the virus into the central nervous system (mechanism described for SARS CoV-1).

ELIGIBILITY:
Inclusion Criteria:

* - adult (≥ 18 years old, unprotected);
* for COVID-19 + patients: COVID-19 + diagnosis; with quantitative or qualitative anomalies in taste and smell; first symptoms appeared in less than 21 days
* for healthy subjects: have never presented any sign of COVID ; confirmed by recent negative serology
* understanding French;
* affiliated to social security;
* having a BMI between 20 and 30;
* preferably non-smokers and in the event of recruitment difficulties, smokers but with smoking <5 packs - year
* signature of the informed consent form

Exclusion Criteria:

* respiratory signs or symptoms (rhinitis, cough, shortness of breath at rest);
* temperature above 37.5 ° C;
* existence of a chronic respiratory pathology (including asthma and COPD in the first row);
* pregnant women ;
* protected minors and adults, persons deprived of their liberty;
* not affiliated to a social security (including AME);
* contraindication to MRI (pace maker, intracranial implants, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Intensity of the emotional response to hypoxic exposure (14.3 et 12.7% FIO2) | 10 minutes
  Slope of the relation between the intensity of a hypoxic stimulus to the intensity of the emotional response (visual analog scale, VAS : 0 is no pain and 10 is the worst pain)

SECONDARY OUTCOMES:
Perception of a hypoxic stimulus induced dyspnea (14.3 et 12.7% FIO2) | 5 minutes
  ratings of dyspnea immediately after a hypoxic stimulus: Multidisciplinary Dyspnea Profile, MDP : 0 is no change and 10 is unbearable
Perception of a hypercapnic stimulus induced dyspnea (7% CO2) | 10 minutes
  ratings of dyspnea intensity and unpleasantness during a hypercapnic stimulus (visual analog scale, VAS : 0 is no pain and 10 is the worst pain)
Perception of a hypercapnic stimulus induced dyspnea (7% CO2) | 5 minutes
  ratings of dyspnea immediately after a hypercapnic stimulus: Multidisciplinary Dyspnea Profile, MDP : 0 is no change and 10 is unbearable
Perception of a inspiratory mechanical constraint induced dyspnea | 10 min
  ratings of dyspnea intensity and unpleasantness during an inspiratory mechanical constraint (visual analog scale, VAS: 0 is no pain and 10 is the worst pain)
Perception of a inspiratory mechanical constraint induced dyspnea | 5 minutes
  ratings of dyspnea immediately after an inspiratory mechanical constraint induced dyspnea(Multidisciplinary Dyspnea Profile, MDP: 0 is no change and 10 is unbearable)
brain MRI | 1,5 hours
  Multimodal MRI (including anatomical MRI, resting-state functional MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- Département R3S, hôpital de la pitié-salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No